CLINICAL TRIAL: NCT04008238
Title: Prospective Identification of Predictive Biomarkers of Trabectedin Efficacy in Non-L Soft-tissue Sarcoma Patients
Acronym: PIPER
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Bergonié (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: IB 2019-02; 2019-A02137-50 (Other: ID-RCB)
Record Dates: First submitted 2019-07-02; First posted 2019-07-05 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-10

CONDITIONS: Soft Tissue Sarcoma Adult; Undifferentiated Pleomorphic Sarcoma; Epithelioid Sarcoma; Solitary Fibrous Tumors; Hemangioendothelioma; Desmoplastic Round Cell Tumor; Synovial Sarcoma
Keywords: Soft-tissue sarcoma; Predictive biomarkers; Next-generation sequencing
MeSH Terms: conditions — Histiocytoma, Malignant Fibrous; Sarcoma; Solitary Fibrous Tumors; Hemangioendothelioma; Sarcoma, Synovial | interventions — Trabectedin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Biomarker analysis (Experimental): This study is a single arm study with biomarker analysis
  Interventions: Drug: Trabectedin

INTERVENTIONS:
Drug: Trabectedin — - Trabectedin will be prescribed as per market authorization and will be administered by intraveinous infusion (1,5 mg/m²) every 3 weeks. A treatment cycle is defined as a 3-weeks period

SUMMARY:
This is a biology driven, monocentric study, designed to identify biomarkers of activity of trabectedin in patients with advanced non-L soft-tissue sarcoma. The aim of this study is to implement high-throughput profiling technologies to identify predictive biomarkers of trabectedin efficacy through sequential tumor biopsies and blood sample collection in sarcoma patients.

DETAILED DESCRIPTION:
The identification of predictive biomarkers of the clinical benefit of trabectedin is a crucial issue to identify potential responders particularly for non-L sarcomas. Considering that the molecular profile of STS can change over time, an analysis of archival tumor material may not be a reliable method to identify predictive biomarkers of response, and thus high-throughput technologies may be promising to identify STS markers for prediction of response to trabectedin. For study purpose, blood and tumor samples will be obtained for genetic and immunological profiling at baseline, during treatment by trabectedin and at disease progression.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years,
2. Histology: undifferentiated pleomorphic sarcomas, epithelioid sarcomas, solitary fibrous tumors, hemangioendothelioma, desmoplastic round cell tumors, synovial sarcomas or other non-leiomyosarcoma/non-liposarcoma softtissue sarcoma. As per the Frech NCI recommendation, diagnosis must be reviewed or confirmed by the RRePS Network (Réseau de Référence en Pathologie des Sarcomes des tissus mous et des Viscères),
3. Locally advanced/unresectable and/or metastatic disease,
4. Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2 (Appendix 1),
5. Measurable disease according to RECIST v1.1,
6. Indication of trabectedin according to market authorization,
7. At least one target lesion that can be biopsied for research,
8. Women of childbearing potential must have a negative serum pregnancy test before study entry,
9. Patient with a social security in compliance with the French law,
10. Voluntary signed and dated written informed consent prior to any study specific procedure,
11. Women must agree to use a medically acceptable method of contraception throughout the treatment period and for 3 months after discontinuation of trabectedin. Men must agree to use a medically acceptable method of contraception throughout the treatment period and for 5 months after discontinuation of trabectedin. Subjects of childbearing potential are those who have not been surgically sterilized or have not been free from menses for >=1 year.

Exclusion Criteria:

1. Previous treatment with trabectedin,
2. Known hypersensitivity to any of its components,
3. Patients with an active serious or uncontrolled infection upon investigator judgement,
4. Radiological evidence of symptomatic or progressive brain metastases,
5. Abnormal coagulation contraindicating biopsy,
6. Any medical and/or biological contra-indication to treatment by trabectedin as per market authorization specification (as per investigator judgement),
7. Patients unable to receive corticotherapy,
8. Previous or current malignancies of other histologies within the last 2 years, with the exception of in situ carcinoma of the cervix, and adequately treated basal cell or squamous cell carcinoma of the skin and prostate cancer,
9. Evidence of severe or uncontrolled systemic disease (uncontrolled hypertension, active bleeding diatheses, or active Hepatitis B, C and HIV),
10. Any condition which in the Investigator's opinion makes it undesirable for the subject to participate in the trial or which would jeopardize compliance with the protocol,
11. Individuals deprived of liberty or placed under guardianship,
12. Pregnant or breast feeding women,
13. Previous enrolment in the present study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2020-01-06 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Efficacy of trabectedin: objective response [OR] or stable disease [SD] > 6 months | Throughout the treatment period, an expected average of 6 months
  Efficacy of trabectedin is defined as objective response [OR] or stable disease [SD] > 6 months. Absence of efficacy is defined as progressive disease [PD] within 2 months.

SECONDARY OUTCOMES:
Safety profile of trabectedin: Common Terminology Criteria for Adverse Events version 5 | Throughout the treatment period, an expected average of 6 months
  Toxicity graded using the Common Terminology Criteria for Adverse Events version 5.
Safety profile of biopsy: Common Terminology Criteria for Adverse Events version 5 | Throughout the treatment period, an expected average of 6 months
  Toxicity graded using the Common Terminology Criteria for Adverse Events version 5.

CONTACTS AND LOCATIONS:
Locations (1):
- Institut Bergonie, Bordeaux, France

IPD SHARING:
Plan to Share IPD: No